CLINICAL TRIAL: NCT00122772
Title: CRP on Radiobiological and Clinical Studies on Viral-induced Cancer's Response to Radiotherapy With Comprehensive Morbidity Assessment
Brief Title: CRP on Radiobiological and Clinical Studies on Viral-Induced Cancer's Response to Radiotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33026
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- EBR plus 2 HDBT fractions (Experimental): External Beam Radiotherapy High Dose Brachytherapy (2 fractions of 9Gy)
  Interventions: Radiation: Radiotherapy
- EBR plus 4 fractions HDBT (Active Comparator): External Beam Radiotherapy High Dose Brachytherapy (4 fractions of 7Gy)
  Interventions: Radiation: Radiotherapy
- EBR/2 HDBT fractions/Chemotherapy (Experimental): External Beam Radiation
  High Dose Brachytherapy (2 fractions of 9Gy)
  Cisplatin
  Interventions: Radiation: Radiotherapy/Cisplatin
- EBR/4 fractions HDBT/chemotherapy (Experimental): External Beam Radiation
  High Dose Brachytherapy (4 fractions of 7Gy)
  Cisplatin
  Interventions: Radiation: Radiotherapy/Cisplatin

INTERVENTIONS:
Radiation: Radiotherapy — External Beam Radiation 46Gy in 23 daily fractions
  High Dose Brachytherapy 2 fractions of 9Gy
  Arms: EBR plus 2 HDBT fractions
Radiation: Radiotherapy — External Beam Radiotherapy 46Gy in 23 daily fractions
  High Dose Brachytherapy 4 fractions of 7Gy
  Arms: EBR plus 4 fractions HDBT
Radiation: Radiotherapy/Cisplatin — External Beam Radiation 46Gy in 23 daily fractions
  High Dose Brachytherapy 2 fractions of 9Gy
  Cisplatin 40 mg/sqm weekly
  Arms: EBR/2 HDBT fractions/Chemotherapy
Radiation: Radiotherapy/Cisplatin — External Beam Radiotherapy 46Gy in 23 daily fractions
  High Dose Brachytherapy 4 fractions of 7Gy
  Cisplatin 40mg/sqm weekly
  Arms: EBR/4 fractions HDBT/chemotherapy

SUMMARY:
The purpose of this trial is to study clinical effects of two/four high dose rate (HDR) brachytherapy applications and teletherapy with or without weekly cisplatin in cervix cancer.

DETAILED DESCRIPTION:
This study uses 2x2 design to test external beam radiotherapy (46 Gy in 23 daily fractions) with and without HDR brachytherapy (2 fractions of 9 Gy versus 4 fractions of 7 Gy) with and without weekly Cisplatin (40 mg/sqm) The overall objective was to test the clinical outcome and toxicity of a resource-sparing schedule of radiotherapy with or without chemotherapy treatment for cervix cancer, to detect molecular markers that will predict tumor control/resistance and to establish whether E6 and E7 viral proteins predict cellular radiosensitivity in oxic and hypoxic conditions in vitro and tumor control/resistance in vivo. A new component of the CRP was added, for which the objective is to optimize the data capture, provide more details of normal tissue outcomes following cancer treatments in developing countries and validate this approach using patients participating in the ongoing CRP. This will be achieved by exploring data capture using the questionnaire template on a computer in face-to-face interviews ("active" data collection) and comparing it with standard data collection obtained from the clinical notes ("passive" data collection) during the still ongoing CRP E3.30.24. The method of data collection will be chosen at random for each case stratified by centre. The reason for using an ongoing CRP is that it will test the usefulness of the new method and validate it in a multicentre study. During the performance of the new CRP, the same institutions as for E3.30.24 will be engaged.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically confirmed cervix cancer.
* FIGO stage IIB and IIIB
* Age over 18 years
* Karnofsky status >/= 50
* No significant medical contraindications to the administration of full dose chemotherapy.
* Adequate bone marrow function -- Haemoglobin ³ 10 g/dl without or with transfusion, white blood count ³ 4000/mL, platelet count ³ 140,000/mL.
* Adequate renal function: creatinine < 1.2 mg/dL or 120 μmol/l (urinary diversion is permitted). Electrolytes and calcium within normal limits for institution. Liver function tests if clinically indicated. Tests have to be obtained within 30 days before registration.
* Expected good compliance for follow-up.
* Written informed consent for participation in this study.

EXCLUSION CRITERIA:

* Recent malignancy, other than the index cervical carcinoma or non-melanoma cutaneous cancers, diagnosed within 5 years of entry
* Life expectancy <6 months, for any reason other than the index cervical carcinoma
* Any severe medical ailment, continuing pregnancy, or breast feeding, as conditions that interfere in present treatment
* Previous chemotherapy in past 1 year
* Severe psychiatric disorder, making compliance and follow-up difficult.
* Paraaortic nodes (PAN >1 cm), suspicious or positive for metastatic involvement on radiological imaging. (Note: patients with positive pelvic lymph nodes are still eligible for the study, but they cannot have suspicious or positive PAN.)
* Bilateral hydronephrosis
* Prior radiation to the pelvis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2005-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome | 5 years
Treatment Toxicity | 3 months
Molecular markers that will predict tumor control/resistance | 5 years
Whether E6 and E7 viral proteins predict cellular radiosensitivity in oxic and hypoxic conditions in vitro and tumor control/resistance in vivo | 5 years
Effectiveness of a questionnaire template on a computer in face-to-face interviews in a multicentre multinational study. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo H. Zubizarreta, M.D., Study Director — International Atomic Energy Agency (IAEA)
Locations (11):
- University of Vienna; Department of Radiotherapy and Radiobiology, Vienna, Austria
- rmandade de Santa Casa de Misericordia de Porto Alegre; Hospital Santa Rita, Porto Alegre, Brazil
- Peel Regional Cancer Centre, Mississauga, Ontario, Canada
- Department of Atomic Energy (DAE); Tata Memorial Centre (TMC); Tata, Mumbai, India
- Institut National d'Oncologie, Rabat, Morocco
- Radiotherapy and Oncology University Clinic, Skopje, North Macedonia
- Bahawalpur Institute of Nuclear Medicine and Oncology (BINO), Bahawalpur, Pakistan
- Instituto Nacional de Enfermedades Neoplásicas, Lima, Peru
- Department of Radiation Oncology, Groote Schuur Hospital, Cape Town, South Africa
- National Cancer Center, Seoul, South Korea
- Christie Hospital; NHS Trust, Manchester, United Kingdom

REFERENCES:
- [Background] Nag S, Chao C, Erickson B, Fowler J, Gupta N, Martinez A, Thomadsen B; American Brachytherapy Society. The American Brachytherapy Society recommendations for low-dose-rate brachytherapy for carcinoma of the cervix. Int J Radiat Oncol Biol Phys. 2002 Jan 1;52(1):33-48. doi: 10.1016/s0360-3016(01)01755-2. PMID 11777620
- [Background] Nag S, Erickson B, Thomadsen B, Orton C, Demanes JD, Petereit D. The American Brachytherapy Society recommendations for high-dose-rate brachytherapy for carcinoma of the cervix. Int J Radiat Oncol Biol Phys. 2000 Aug 1;48(1):201-11. doi: 10.1016/s0360-3016(00)00497-1. PMID 10924990
- [Background] Petereit DG, Pearcey R. Literature analysis of high dose rate brachytherapy fractionation schedules in the treatment of cervical cancer: is there an optimal fractionation schedule? Int J Radiat Oncol Biol Phys. 1999 Jan 15;43(2):359-66. doi: 10.1016/s0360-3016(98)00387-3. PMID 10030262
- [Background] Whitney CW, Sause W, Bundy BN, Malfetano JH, Hannigan EV, Fowler WC Jr, Clarke-Pearson DL, Liao SY. Randomized comparison of fluorouracil plus cisplatin versus hydroxyurea as an adjunct to radiation therapy in stage IIB-IVA carcinoma of the cervix with negative para-aortic lymph nodes: a Gynecologic Oncology Group and Southwest Oncology Group study. J Clin Oncol. 1999 May;17(5):1339-48. doi: 10.1200/JCO.1999.17.5.1339. PMID 10334517
- [Background] Morris M, Eifel PJ, Lu J, Grigsby PW, Levenback C, Stevens RE, Rotman M, Gershenson DM, Mutch DG. Pelvic radiation with concurrent chemotherapy compared with pelvic and para-aortic radiation for high-risk cervical cancer. N Engl J Med. 1999 Apr 15;340(15):1137-43. doi: 10.1056/NEJM199904153401501. PMID 10202164
- [Background] Green JA, Kirwan JM, Tierney JF, Symonds P, Fresco L, Collingwood M, Williams CJ. Survival and recurrence after concomitant chemotherapy and radiotherapy for cancer of the uterine cervix: a systematic review and meta-analysis. Lancet. 2001 Sep 8;358(9284):781-6. doi: 10.1016/S0140-6736(01)05965-7. PMID 11564482
- [Background] Pearcey R, Brundage M, Drouin P, Jeffrey J, Johnston D, Lukka H, MacLean G, Souhami L, Stuart G, Tu D. Phase III trial comparing radical radiotherapy with and without cisplatin chemotherapy in patients with advanced squamous cell cancer of the cervix. J Clin Oncol. 2002 Feb 15;20(4):966-72. doi: 10.1200/JCO.2002.20.4.966. PMID 11844818
- See also: International Atomic Energy Agency, Research Contracts Administration — http://www.iaea.org